CLINICAL TRIAL: NCT06089876
Title: The Use of Step Tracker Mobile Applications in Overweight and Obese Adolescents for the Promotion of Physical Activity and the Improvement of Kinanthropometric Variables, Fitness and Psychological State
Brief Title: The Use of Mobile Applications in Obese and Overweight Adolescents for Health Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Raquel Vaquero-Cristóbal, Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFYNNTT-ESOCARM
Record Dates: First submitted 2023-10-05; First posted 2023-10-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Overweight Adolescents; Obesity, Adolescent; Physical Inactivity; Mobile Phone Use; Behavior, Health
MeSH Terms: conditions — Pediatric Obesity; Sedentary Behavior; Cell Phone Use; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Strava" Application (Experimental): STRAVA is an application that allows you to record your physical activity. Using GPS, it allows you to record the distance traveled with different types of physical activity (walking, running, swimming, among others). In addition, it allows you to create a community and clubs within the same community with which you can propose group trails.
  Interventions: Behavioral: STRAVA mobile application
- Control Group (No Intervention): They will not use any type of sports technology application. They will continue to perform their daily activities without intervention.

INTERVENTIONS:
Behavioral: STRAVA mobile application — The adolescents in the intervention group will use the STRAVA mobile application for a period of 10 weeks. To do so, they will follow the instructions provided by the researchers on the frequency of use, the distance to be covered and how to record it.
  Arms: "Strava" Application

SUMMARY:
Overweight and obesity, understood as an accumulation of abnormal and excessive fat, are the second leading cause of preventable and avoidable mortality in developed countries, with more than 340 million children and adolescents affected by this disease worldwide. As a consequence, overweight and obesity at an early age is already considered a pandemic by the World Health Organization (WHO), with a high incidence in developed countries.

The abuse of new technologies has remained at worrying levels in the post-COVID period, favoring an increase in the adolescent population considered sedentary. In this regard, up to 70% of adolescents show sedentary behaviors, especially affecting the time spent on screens by both males (93.8%) and females (87.2%). Thus, the use of the cell phone has been shown to be a determining factor, since between 10% and 16% of adolescents show a problematic use of this device, affecting, among other aspects, their behavior during their free time.

In recent years there has been an increase in sedentary time among adolescents and a decrease in the practice of physical activity that has favored a greater accumulation of body fat and increased the probability of being overweight or obese. In this context, some studies have tried to encourage the practice of physical activity in the school context in overweight and obese population, being these interventions effective to improve body composition.

However, these interventions also have their detractors, who argue that the hours of Physical Education are too limited to dedicate so much time to a single content, and that the pedagogical component is often overlooked in their implementation. As an alternative to the above, it has been suggested that Physical Education classes could be used to promote interventions that encourage adolescents to practice physical activity in their free time, and mobile applications could be used to monitor the activity carried out by adolescents, but also as an element that generates adherence and enjoyment in this population. Research in this population using these technologies is scarce, therefore, this project aims to determine the effectiveness of a ten-week intervention promoted from the subject of physical education in which a mobile application is used after school hours on physical activity, body composition and fitness in overweight or obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Be a student of compulsory secondary education
* Present an BMI > 25.0
* Not present any disease or surgical operation that would prevent the performance of the physical tests or the follow-up of the established intervention.
* Complete the questionnaires provided and carry out the established tests in their entirety.
* Have access to any mobile device that allows access to the technological sports applications used in the intervention.

Exclusion Criteria:

* Failure to complete the questionnaires provided and/or to take the prescribed tests in their entirety.
* Failure to complete scheduled intervention activities.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-02-16 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Level | Through study completion, an average of 25 weeks
  The level of physical activity was measured using the Spanish version of the physical activity questionnaire for adolescents (PAQ-A). This questionnaire is composed of nine items, the first eight of which are completed on a Likert scale of 1 to 5 points. The arithmetic mean of the scores of the first eight items provides a final physical activity score. The minimum score ranges from 1 to 5 points. A 1 indicates that the level of physical activity of adolescents is very low, while a 5 indicates that the level of physical activity is very high.
Use of internet | Through study completion, an average of 25 weeks
  The Questionnaire of Experiences Related to Internet Use (CERI) will be used to analyze problematic Internet use by adolescents. This instrument is composed of 10 items that are completed on a Likert scale from 1 to 4 points (1: never; 4: almost always), with the sum of the 10 items being the final score of the questionnaire. The questionnaire indicates problematic use (PU), when the score is higher than 26 in the CERI; occasional problems (OP), when the score is between 18 and 25 in the CERI; and no problems (NP), when the score is lower than 18 in the CERI. It has been previously validated and has a Cronbach's alpha of 0.77 for CERI.
Use of mobile phone | Through study completion, an average of 25 weeks
  The Questionnaire of Experiences Related to Mobile Phones (CERM) will be used to analyze problematic mobile phone use by adolescents. This instrument is composed of 10 items that are completed on a Likert scale from 1 to 4 points (1: never; 4: almost always), with the sum of the 10 items being the final score of the questionnaire. The questionnaire indicates problematic use (PU), when the score is higher than 24 in the CERM; occasional problems (OP), when the score is between 16 and 23 in the CERM; and no problems (NP), when the score is lower than 16 in the CERM. It has been previously validated and has a Cronbach's alpha of 0.80 for CERM.
Handgrip Strength | Through study completion, an average of 25 weeks
  To assess upper limb strength, participants will be instructed to utilize a Takei Tkk5401 digital handheld dynamometer (Takei Scientific Instruments, Tokyo, Japan) and squeeze it with their elbow fully extended. This position is chosen because it allows for maximum force production.
VO2 max. | Through study completion, an average of 25 weeks
  To assess the cardiorespiratory capacity of adolescents, the 20-m shuttle run test, an incremental test of high validity and reliability for use with adolescents, will be used. Using the formula of Léger and the speed at which the subject finishes the test, maximal oxygen consumption (VO2 max) is predicted.
Countermovement jump (CMJ) | Through study completion, an average of 25 weeks
  For the CMJ, a force platform with a sampling frequency of 200 Hz (MuscleLab, Stathelle, Norway) will be used. During the CMJ test, participants will be instructed to execute a maximal vertical jump while keeping their hands on their waists and ensuring full trunk extension throughout the flight phase.
Hamstrings flexibility | Through study completion, an average of 25 weeks
  To measure hamstring and lumbar flexibility, the sit-and-reach test will be used. The adolescents have to perform maximum trunk flexion, keeping their hands and knees fully extended, to reach the maximum possible distance by sliding their palms, one on top of the other, across the box.
Speed | Through study completion, an average of 25 weeks
  To measure speed, the 20-m sprint will be used, in which adolescents, starting from a standing position behind a line, and initiating the run at a time of their choice, must cover 20 m in the shortest possible time. Single-beam photocells (Polifemo Light; Microgate, Italy) placed at hip height will be used for the measurement.
Curl-up | Through study completion, an average of 25 weeks
  To assess abdominal muscle endurance will be use Curl-up. The highest number of repetitions the subject completes in one minute will be recorded.
Push-up | Through study completion, an average of 25 weeks
  To assess upper limb strength will be used Push-up test. The subject will perform as many repetitions as possible in one minute, or until reaching exhaustion (Castro-Piñero et al., 2010).
Height | Through study completion, an average of 25 weeks
  To measure height, a SECA measuring rod should be used. Adolescents should stand barefoot with their backs against the measuring rod, heels of their feet together and their gaze straight ahead. Measurements will be obtained in centimeters and will be repeated 2 times for each subject. A third measurement will only be taken if the difference between the first and second measurement is greater than 1%.
Weight | Through study completion, an average of 25 weeks
  A Tanita BC 418-MA Segmental scale (Tanita, Tokyo) will be used to measure body weight. The subject will step on the scale with both feet inside the scale and looking straight ahead, without leaning the body. Values will be obtained in kilograms and two measurements will be carried out on each subject. If the difference between both measurements is greater than 1%, a third measurement will be taken
Fat mass | Through study completion, an average of 25 weeks
  To obtain the fat mass, it will be necessary to previously measure the triceps, thigh and leg folds, and the waist, hip, relaxed arm, thigh and leg perimeters. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the fat mass can be calculated using the formula of Slaughter.
Fat-free mass | Through study completion, an average of 25 weeks
  To obtain the fat-free mass, it will be necessary to previously measure the triceps, thigh and leg folds, and the perimeters of the waist, hip, relaxed arm, thigh and leg. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the-fat free mass can be calculated using the formula of Poortmans.
BMI | Through study completion, an average of 25 weeks
  Previously obtained height and weight measurements will be used to establish the BMI. The formula used will be weight/height^2, and the result will be obtained in kg/m^2. This index is commonly used and is related to metabolic and cardiovascular diseases in adolescents and adults.

SECONDARY OUTCOMES:
User version of the Mobile Application Rating Scale | Through study completion, an average of 25 weeks
  The User version of the Mobile Application Rating Scale (uMARS) is a scale consisting of 26 items completed using a Likert scale ranging from 1 to 5 points. This scale allows for the assessment of 6 dimensions, which include engagement, functionality, aesthetics, information, subjective quality, and perceived impact of the mobile application. Engagement scores range between 5 and 25 points; functionality and information between 4 and 20; aesthetics between 3 and 15; subjective quality between 4 and 20; and perceived impact between 6 and 30. A higher score in all cases indicates a better assessment of the app.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vaquero-Cristóbal, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mateo-Orcajada A, Ponce-Ramirez CM, Abenza-Cano L, Vaquero-Cristobal R. Effects of 10 Weeks of Walking With Mobile Step-Tracking Apps on Body Composition, Fitness, and Psychological State in Adolescents Who Are Overweight and Obese: Randomized Controlled Trial. J Med Internet Res. 2024 Dec 10;26:e55243. doi: 10.2196/55243. PMID 39656510